CLINICAL TRIAL: NCT06237764
Title: Genetic and Risk Factors in Exfoliation Glaucoma Patients in Sweden
Brief Title: Genetic and Risk Factors in Exfoliation Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: Glaugene1
Record Dates: First submitted 2024-01-06; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Glaucoma Capsulare; Genetic Predisposition to Disease; Risk Reduction
Keywords: Glaucoma; Exfoliation; Risk factors; Genetics
MeSH Terms: conditions — Exfoliation Syndrome; Genetic Predisposition to Disease; Risk Reduction Behavior; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genetics in exfoliation glaucoma: Prospective recruited patients suffering from exfoliation glaucoma.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
Prospective non-randomised cohort study enrolling patients with exfoliation glaucoma. All patients were ophthalmological examined at inclusion. Blood samples were taken for genetic analysis.

DETAILED DESCRIPTION:
Patients & examinations In this prospective non-randomised cohort study, the investigators enrolled patients with exfoliation glaucoma at the Ophthalmology Department of the Skaraborg's Hospital, Skövde, and Sahlgrenska University Hospital, Gothenburg, from 1st January, 2014, to 31st December, 2017. All patients were followed-up for three years ± three months. Informed consent was obtained from all patients. The study protocol was granted ethical approval by the University of Gothenburg (DN:119-12). The study was performed in accordance with the tenets of the Declaration of Helsinki.

At the recruiting visit, an ophthalmic nurse checked the visual acuity of patients with a Snellen's chart and performed a visual field test. Humphrey Field Analysis was performed using the software threshold 24-2. Subsequently, an ophthalmologist measured the intracoular pressure (IOP) with a Goldmann applanation tonometer and performed slit-lamp biomicroscopy, including gonioscopy. Pupils were then dilated with 2.5% phenylephrine and 0.5% tropicamide. After 20 min, the presence of exfoliation was confirmed, and the optic nerve was assessed using a 90-D lens. Subsequently, the central corneal thickness (CCT) was measured using an ultrasound device. The average value of seven measurements was automatically calculated. At the end of the visit, blood samples were collected. The number of medicines was registered as the number of compounds and not the number of bottles used.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of exfoliation glaucoma based on the criteria established by the European Glaucoma Society Terminology and Guidelines for Glaucoma, i.e., an untreated IOP of ≥21 mmHg, an open anterior chamber angle, glaucomatous visual field defects (at least two repeatable Humphrey 24-2 tests), glaucomatous optic nerve damage, and the presence of exfoliation material.
* Patients must performed at least five reliable visual field tests during the 3-year follow-up, with reliability defined as false positives ≤15%, false negatives ≤20%, and/or fixation losses ≤30%.
* Age ≤85 years at the recruiting visit.

Exclusion Criteria:

* A diagnosis of advanced glaucoma defined as mean deviation (MD) ≥18 decibel (dB) and/or visual field index (VFI) ≤40% because of 'floor effects,' in which further loss of visual field defects can no longer be detected.
* History of glaucoma surgery other than uneventful cataract surgery or selective laser trabeculoplasty (SLT).
* Other eye diseases (central venous occlusion, retinal detachment, etc.) that could affect the visual fields during the 3-year follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this prospective non-randomised cohort study, the investigators enrolled patients with exfoliation glaucoma at the Ophthalmology Department of the Skaraborg's Hospital, Skövde, and Sahlgrenska University Hospital, Gothenburg.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Visual field progression using mean deviation (MD) | At least three years follow-up
  The visual field progression was studied with three methods. The first method was based on MD visual field. The difference in MD values from the beginning to the end of the study was calculated. Higher values indicated higher progression. Results will be analyzed using linear regression.
Visual field progression using visual field index (VFI) | At least three years follow-up
  The second method was based on VFI. A device calculated the VFI and performed a regression analysis to calculate the rate of progression (ROP). The machine calculated the ROP as the amount of VFI deterioration (%)/year. The ROP calculation is also referred to as a 'trend analysis.' Results will be analyzed using linear regression.
Visual field progression using the guided progression analysis (GPA) strategy | At least three years follow-up
  The third method was the GPA, which is also included in the device and performed automatically (GPA Alert) but differs from ROP. GPA is an 'event analysis,' while ROP is a 'trend analysis'. The machine compares every single point before examinations. The GPA alert result options for progression are 'no', 'possible', and 'likely'. We evaluated glaucoma as 'no progression' or 'progression', the latter including both 'possible' and 'likely'. Results will be analyzed using logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Ayala, MD/PhD, Principal Investigator — Göteborg University
Locations (1):
- Skaraborg Hospital, Skövde, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Ground information of the cohort like age, sex, genetic analysis, risk factors, etc.
Supporting Information: Study Protocol, SAP
Time Frame: Data already available upon request until the end of 2026.
Access Criteria: Other researchers working with exfoliation glaucoma patients.

REFERENCES:
- [Result] Ayala M, Zetterberg M, Zettergren A. Single nucleotide polymorphisms in LOXL1 as biomarkers for progression of exfoliation glaucoma in Sweden. Acta Ophthalmol. 2023 Aug;101(5):521-529. doi: 10.1111/aos.15630. Epub 2022 Dec 23. PMID 36564963

DOCUMENTS (2):
  • Study Protocol (2012-05-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT06237764/Prot_000.pdf
  • Statistical Analysis Plan (2012-05-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT06237764/SAP_001.pdf